CLINICAL TRIAL: NCT02045693
Title: A Phase1, Open-Label, Drug-Drug Interaction Study Between Methadone and Daclatasvir/Asunaprevir/BMS-791325 3 DAA FDC + 75mg BMS-791325 and Between Buprenorphine/Naloxone and Daclatasvir/Asunaprevir/BMS-791325 3 DAA FDC +75mg BMS-791325
Brief Title: Drug Interaction & Methadone & Buprenorphine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: AI443-108
Record Dates: First submitted 2014-01-21; First posted 2014-01-27 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Methadone; 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide; Buprenorphine; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: Methadone + DCV 3DAA FDC + BMS-791325 (Experimental): Methadone 40-120 mg tablet or solution orally once on Day 1
  Methadone 40-120 mg tablet or solution orally once daily + DCV 3DAA FDC (Daclatasvir 30 mg/Asunaprevir 200 mg/BMS-791325 75 mg 3 direct-acting antiviral (3DAA) fixed dose combination tablet) orally twice daily + BMS-791325 75 mg tablet orally twice daily on Days 2 through 12
  Interventions: Drug: Methadone; Drug: DCV 3DAA FDC; Drug: BMS-791325
- Part 2: Buprenorphine/Naloxone + DCV 3DAA FDC + BMS-791325 (Active Comparator): Buprenorphine/Naloxone 8/2 - 24/6 mg tablet or sublingual film orally once on Day 1
  Buprenorphine/Naloxone 8/2 - 24/6 mg tablet or sublingual film orally once + DCV 3DAA FDC (Daclatasvir 30 mg/Asunaprevir 200 mg/BMS-791325 75 mg 3DAA fixed dose combination tablet) orally twice daily + BMS-791325 75 mg tablet orally twice daily on Days 2 through 12
  Interventions: Drug: DCV 3DAA FDC; Drug: BMS-791325; Drug: Buprenorphine; Drug: Naloxone

INTERVENTIONS:
Drug: Methadone
  Arms: Part 1: Methadone + DCV 3DAA FDC + BMS-791325
Drug: DCV 3DAA FDC
Drug: BMS-791325
Drug: Buprenorphine
  Arms: Part 2: Buprenorphine/Naloxone + DCV 3DAA FDC + BMS-791325
Drug: Naloxone
  Arms: Part 2: Buprenorphine/Naloxone + DCV 3DAA FDC + BMS-791325

SUMMARY:
The purpose of this study is to assess the effects of steady state DCV/ASV/BMS-791325 fixed dose combination (FDC) + 75mg BMS-791325 on the Pharmacokinetics (PK) of Methadone in subjects with the stable dose of Methadone and on the PK of Buprenorphine in subjects with the stable dose of Buprenorphine.

DETAILED DESCRIPTION:
IND number: 101,943

Primary purpose: Other: Phase 1 Clinical Pharmacology drug interaction study in healthy subjects

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subject must be on stable Methadone or Buprenorphine regimens for at least 28 days prior to screening

Exclusion Criteria:

* Subjects must be healthy except for history of Methadone or Buprenorphine treatment regimens
* Prior exposure to DCV, ASV or BMS-791325 within 3 months of screening or any other investigational drug or placebo within 4 weeks of study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of R-Methadone for Part 1 | 24 timepoints up to Day 13
Area under the concentration-time curve in one dosing interval (AUC(TAU)) of R-Methadone for Part 1 | 24 timepoints up to Day 13
Cmax of Buprenorphine and Norbuprenorphine for Part 2 | 24 timepoints up to Day 13
AUC(TAU) of Buprenorphine and Norbuprenorphine for Part 2 | 24 timepoints up to Day 13

SECONDARY OUTCOMES:
Cmax of S-Methadone and Total Methadone for Part 1 | 24 timepoints up to 13 days
AUC(TAU) of S-Methadone and Total Methadone for Part 1 | 24 timepoints up to 13 days
Concentration at 24 hours (C24) of S-Methadone, Total Methadone and R-Methadone for Part 1 | 24 timepoints up to 13 days
Time of maximum observed concentration (Tmax) of S-Methadone, Total Methadone and R-Methadone for Part 1 | 24 timepoints up to 13 days
C24 of Buprenorphine and Norbuprenorphine for Part 2 | 24 timepoints up to 13 days
Tmax of Buprenorphine and Norbuprenorphine for Part 2 | 24 timepoints up to 13 days
Ratio of metabolite AUC(TAU) to parent AUC(TAU) (MR_AUC(TAU)) of Norbuprenorphine to Buprenorphine | 24 timepoints up to 13 days
Cmax of of Daclatasvir (DCV) , Asunaprevir (ASV) , BMS-791325, and BMS-794712 | 10 timepoints on Day 12
AUC(TAU) of DCV, ASV, BMS-791325, and BMS-794712 | 10 timepoints on Day 12
Concentration at 12 hours (C12) of DCV, ASV, BMS-791325, and BMS-794712 | 10 timepoints on Day 12
Tmax of DCV, ASV, BMS-791325, and BMS-794712 | 10 timepoints on Day 12
MR_AUC(TAU) for BMS-794712 to BMS-791325 | 10 timepoints on Day 12
Incidence of Adverse Events (AEs), Serious Adverse Events (SAEs), death and AEs leading to discontinuation | Up to day 13
Results of vital signs, Electrocardiograms (ECGs), Physical Examinations (PEs) and clinical labs | Up to day 13
Scores of Clinical Opiate Withdrawal Scale (COWS), Subjective Opiate Withdrawal Scale (SOWS), Objective Opiate Withdrawal Scale (OOWS), and Opiate Overdose Assessment (OOA) | Up to day 13

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Anaheim Clinical Trials Llc, Anaheim, California
  - Cri Lifetree, Philadelphia, Pennsylvania
  - Lifetree Clinical Research, Salt Lake City, Utah

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx